CLINICAL TRIAL: NCT06710457
Title: Effect of Erector Spinae Plane Block on Postoperative Nausea and Vomiting in Lumbar Disc Herniation Surgery
Brief Title: Effect of Erector Spinae Plane Block on Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gökhan Erdem, Anesthesiology and Reanimation specialist doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ESP PONV
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia; Pain, Postoperative; Nausea and Vomiting, Postoperative
Keywords: Erector spinae plane block; Postoperative nausea vomiting; Apfel score
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane (ESP) block (Active Comparator): Patients will receive an erector spinae plane (ESP) block in addition to standard medical treatment to prevent PONV and postoperative pain.
  Interventions: Other: ESP
- No Erector spinae plane (ESP) block (Active Comparator): Patients will receive standard medical treatment to prevent PONV and postoperative pain.
  Interventions: Other: No ESP

INTERVENTIONS:
Other: ESP — Patients will receive an erector spinae plane (ESP) block in addition to standard medical treatment to prevent PONV and postoperative pain.
  Arms: Erector spinae plane (ESP) block
Other: No ESP — Patients will receive standard medical treatment to prevent PONV and postoperative pain.
  Arms: No Erector spinae plane (ESP) block

SUMMARY:
This study will investigate the hypothesis that preoperative erector spinae plane (ESP) block will reduce the incidence of postoperative nausea and vomiting (PONV) in patients undergoing elective lumbar disc herniation (LDH) surgery. PONV was defined as the presence of nausea and vomiting within 24 hours postoperatively.

DETAILED DESCRIPTION:
The study will include patients aged 18 years and older, with (American Society of Anesthesiologists) ASA physical status I and II, and scheduled for single-level lumbar disc herniation surgery under general anesthesia. Patient characteristics (age, gender, body mass index, etc.), Apfel score, postoperative nausea and vomiting (PONV) status, intraoperative opioid use requirement, surgical duration, postoperative pain status, rescue analgesic and emetic requirement will be recorded. The primary outcome parameter will be the PONV incidence within the postoperative 24 hours. PONV severity during this period will be assessed using a Likert scale from 0 to 10. PONV will be defined as vomiting, marked nausea (numerical rating scale [NRS] ≥4), and/or need for rescue medication. Patients will be assessed for PONV at 0, 2, 4, 12, and 24 hours using the Likert scale. Nausea and its severity, vomiting attacks, need for intraoperative opioid use, pain and its severity, need for additional analgesics, and administration of antiemetic rescue medication will be evaluated as secondary outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* ASA physical status I to II
* One lumbar disc herniation surgery under general anesthesia

Exclusion Criteria:

* body mass index >35 kg/m²)
* history of drug use
* nausea and vomiting before surgery
* psychiatric disorders
* use of antipsychotic or antiemetic drugs
* severe heart disease
* central nervous system diseases
* vertebrobasilar artery insufficiency
* cytostatic therapy
* vestibular diseases
* renal and/or hepatic dysfunction
* pregnant patients
* presence of bleeding diathesis
* patients in a condition where cooperation cannot be established in the post-operative period (mental retardation etc.)
* patient's refusal to accept the block procedure
* allergy to local anesthetics
* injection site infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
PONV | 24 hours
  The primary outcome of the study was the incidence of postoperative nausea and/or vomiting

SECONDARY OUTCOMES:
Severity of nausea | 24 hours
  The degree of nausea was evaluated using the visual analogue scale (VAS), with 0 indicating no nausea or vomiting and 10 indicating the most severe form of unbearable nausea or vomiting. When the PONV score was greater than 4 or vomiting occurs
11 - point numerical rating scale (NRS) | 24 hours
  11-point numerical rating scale for pain (0='no pain' and 10='worst pain possible pain') were explained.
Rescue antiemetic requirement | 24 hours
  Number of additional antiemetic applications
Rescue analgesic requirement | 24 hours
  Number of additional analgesic applications
intraoperative opioid requirement | intraoperative time
  To maintain the bispectral index (BIS) between 40-60, remifentanil will be initiated and titrated between 0.05-0.25 mcg/kg/min, taking into account a 20% increase in MAP (mean arterial pressure) compared to the initial value and a 15% increase in heart rate compared to the initial value.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erdem G, Kavak Akelma F, Nalbant B, Gokbulut Ozaslan N. Effect of erector spinae plane block on postoperative nausea and vomiting in lumbar disc herniation surgery. Reg Anesth Pain Med. 2025 Jun 30:rapm-2025-106756. doi: 10.1136/rapm-2025-106756. Online ahead of print. PMID 40588358